CLINICAL TRIAL: NCT02503683
Title: A Phase 1/2, Randomized, Single-blind, Placebo-Controlled, Single Ascending Dose and Multiple Dose, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Subcutaneously Administered ALN-AAT in Healthy Adult Subjects and Patients With ZZ Type Alpha-1 Antitrypsin Deficiency Liver Disease
Brief Title: A Study of an Investigational Drug, ALN-AAT, in Healthy Adult Subjects and Patients With ZZ Type Alpha-1 Antitrypsin Deficiency Liver Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Observation of low incidence of asymptomatic, transiently elevated liver enzymes in a subset of study subjects
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-AAT-001
Record Dates: First submitted 2015-07-16; First posted 2015-07-21 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Antitrypsin Deficiency Liver Disease
Keywords: RNAi therapeutic; AAT; Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-AAT (Active Comparator)
  Interventions: Drug: ALN-AAT
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-AAT — Single or multiple doses of ALN-AAT by subcutaneous (sc) injection
  Arms: ALN-AAT
Drug: Sterile Normal Saline (0.9% NaCl) — calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered ALN-AAT in Healthy Adult Subjects and Patients with ZZ Type Alpha-1 Antitrypsin Deficiency Liver Disease.

ELIGIBILITY:
Inclusion Criteria:

* Adequate complete blood counts, liver and renal function.
* 12-lead electrocardiogram (ECG) within normal limits
* Female subjects must be of non-childbearing potential; e.g. post-menopausal or pre-menopausal with surgical sterilization
* Male subjects agree to use appropriate contraception
* Willing to provide written informed consent and willing to comply with study requirements
* Nonsmokers for at least 5 years before screening

Exclusion Criteria:

* Any uncontrolled or serious disease, or any medical or surgical condition, that may interfere with participation in the clinical study and/or put the subject at significant risk
* Received an investigational agent within 90 days before the first dose of study drug or are in follow-up of another clinical study
* Active serious mental illness or psychiatric disorder requiring current pharmacological intervention
* History or evidence of alcohol or drug abuse within 12 months before screening.
* History of intolerance to SC injection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
The safety of ALN-AAT evaluated by the proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs), and AEs leading to study drug discontinuation | Part A (SAD phase): through day 70; Part B (MAD) phase: through Day 154; Part C: through Day 224

SECONDARY OUTCOMES:
Profile of Pharmacokinetics (PK) of ALN-AAT | Part A (SAD) phase: up to 21 days; Part B (MAD) phase: up to 105 days; Part C: up to 161 days
  Cmax, tmax, AUC, t1/2
The effect of ALN-AAT on serum levels of AAT protein | Part A (SAD) phase: through day 70; Part B (MAD) phase: through Day 154; Part C: through Day 224

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Haslett, MD, Study Director — Alnylam Pharmaceuticals
Locations (1):
- Richmond Pharmacology, Ltd., London, United Kingdom